CLINICAL TRIAL: NCT01597128
Title: Feasibility Study of The Use of FLEX HD® Surgical Implant or STRATTICE® Reconstructive Tissue Matrix in The Closure of Abdominal Wall Defects With Component Separation in Clean or Contaminated Cases
Acronym: Flex HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Roth (Other)
Responsible Party: Sponsor-Investigator, John Roth, PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-0080-P6A
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2016-10

CONDITIONS: Hernia Repair With Compartment Syndrome
Keywords: Hernia; human tissue; mesh
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flex HD (Active Comparator): Mesh Type
  Interventions: Device: Flex HD
- Strattice (Active Comparator): Use of a second mesh type
  Interventions: Device: Strattice

INTERVENTIONS:
Device: Flex HD — Flex HD mesh for hernia repair
  Arms: Flex HD
Device: Strattice — Strattice mesh for hernia repair
  Arms: Strattice

SUMMARY:
This study examines the feasibility of using Flex HD® Surgical Implant or STRATTICE® Reconstructive Tissue Matrixin the repair of hernias.

DETAILED DESCRIPTION:
At least 100,000 ventral hernia repairs are performed in the U.S. each year. Recently, biologically-based implants derived from acellular human dermis, porcine small intestinal submucosa, and porcine dermis have been reported in a variety of complex abdominal wall repair procedures. A variety of surgical techniques and implant placement methods have been described, with no one standard technique achieving precedence. Biologic implant reinforcement of a myofascial closure by means of component separation, or at a minimum, where three-layer fascial approximation is not possible, sublay placement (i.e., closure of the posterior rectus sheath under the implant) are described strategies. These techniques allow placement of the implant against an intact fascial layer and may improve implant incorporation into host tissue.

The Musculoskeletal Transplant Foundation (MTF) has manufactured and processed Flex HD Acellular Hydrated Dermis. This acellular dermis is derived from human skin. In complicated ventral hernia repairs, this type of graft tissue is necessary. Flex HD has been shown to reduce operative time, lower operative costs and provides minimal elasticity.

The Musculoskeletal Transplant Foundation (MTF) is a non-profit service organization dedicated to providing quality allograft tissue through a commitment to excellence in education, research, recovery and care for recipients, donors and their families. MTF is a national consortium comprised of academic medical institutions, organ procurement organizations and tissue recovery organizations. From their inception, they have been both donor-focused and surgeon-driven. Since their inception in 1987, MTF has recovered more than 60,000 donors and distributed more than 3 million grafts for transplantation.

The Foundation was established by surgeons and teaching institutions to meet the need for a high quality and consistent allograft supply.

ELIGIBILITY:
Inclusion Criteria:• Have given written Informed Consent

* Be 18-85 years of age (inclusive)
* Patient has a ventral or incisional hernia with at least one of the following characteristics

  * Hernia is at least 6cm in transverse dimension
  * History of 2 or more prior ventral or incisional hernia repairs
  * Active or prior infection of the abdominal wall
  * Enterocutaneous fistula to the anterior abdominal wall
  * Mesh requiring mesh removal which would result in a hernia at least 6cm in transverse dimension
* Patients is scheduled to undergo component separation hernia repair
* Have an ASA Score of 3 or less
* Have a BMI between 20 and 55
* Be a candidate for primary approximation of skin and wound following hernia repair
* Have a life expectancy of at least 2 years

Exclusion Criteria:

* Have loss of abdominal domain such that the operation would be impractical or would adversely effect respiratory or cardiovascular function to an unacceptable degree
* Be a candidate for emergency surgery that would make giving valid Informed Consent impractical
* Be currently taking part in another clinical study that conflicts with the current study
* Have active generalized peritonitis or intraperitoneal sepsis
* Have active necrotizing fasciitis
* Have active abdominal compartment syndrome
* Have active untreated metabolic or systemic illness
* Have known active malignancy present
* Be unable to give valid informed consent or comply with required follow-up schedule
* Suffer from mental capacity sufficiently severe to make informed consent unobtainable

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S Roth, M.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

REFERENCES:
- See also: Musculoskeletal Transplant Foundation — http://www.mtf.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were identified in the Minimally Invasive Surgery Clinic at the University of Kentucky Medical Center. Recruitment started in March of 2011 and ended in May of 2014
Groups:
- Flex HD: Human Acellular Dermal Matrix: Flex HD mesh for hernia repair
- Strattice: Porcine Acellular Dermal Matrix: Strattice mesh for hernia repair
Period: Overall Study
Arm/Group | Flex HD | Strattice
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flex HD | Strattice | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10) | 58 (12) | 58 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 10 | 4 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 16 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35
Smoker [Number; unit: participants] | 10 | 12 | 22
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34 (7) | 34 (6) | 34 (6.3)
With Prior Defect [Number; unit: participants] | 11 | 7 | 18
Number of Participants Who Were Employed Prior to the Hernia Repair [Number; unit: participants] | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Hernia Recurrence
Description: Recurrence of hernia based on physical exam and /or CT scan.
Time Frame: 12 months
Measure: Number; unit: percentage of patients
Arm/Group | Flex HD | Strattice
Number analyzed (Participants) | 18 | 17
percentage of patients | 11 | 12

2. Primary Outcome: Wound Occurrence
Description: superficial or deep wound infection, abscess, seroma, cellulitis, necrosis, hematoma or wound dehiscence.
Time Frame: 12 months
Measure: Number; unit: percentage of patients
Arm/Group | Flex HD | Strattice
Number analyzed (Participants) | 18 | 17
percentage of patients | 17 | 29

3. Primary Outcome: Wound Occurrence: Deep Wound Infection
Time Frame: 12 Months
Measure: Number; unit: percentage of patients
Arm/Group | Flex HD | Strattice
Number analyzed (Participants) | 18 | 17
percentage of patients | 0 | 6

4. Primary Outcome: Wound Occurrence: Wound Abscess
Time Frame: 12 Months
Measure: Number; unit: percentage of patients
Arm/Group | Flex HD | Strattice
Number analyzed (Participants) | 18 | 17
percentage of patients | 11 | 18

5. Primary Outcome: Wound Occurrence: Wound Seroma
Time Frame: 12 Months
Measure: Number; unit: percentage of patients
Arm/Group | Flex HD | Strattice
Number analyzed (Participants) | 18 | 17
percentage of patients | 11 | 12

6. Primary Outcome: Wound Occurrence: Wound Cellulitis
Time Frame: 12 Months
Measure: Number; unit: percentage of patients
Arm/Group | Flex HD | Strattice
Number analyzed (Participants) | 18 | 17
percentage of patients | 0 | 6

7. Primary Outcome: Wound Occurrence: Wound Dehiscence
Time Frame: 12 Months
Measure: Number; unit: percentage of patients
Arm/Group | Flex HD | Strattice
Number analyzed (Participants) | 18 | 17
percentage of patients | 11 | 0

8. Primary Outcome: Wound Occurrence: Superficial Wound Infection
Description: Superficial wound infection
Time Frame: 12 months
Measure: Number; unit: percent of patients
Arm/Group | Flex HD | Strattice
Number analyzed (Participants) | 18 | 17
percent of patients | 17 | 29

9. Primary Outcome: Change in SF12 Physical Component Score Between Pre-operation and 12 Months Post-operation
Description: Change in SF12 Physical Component Score from pre-operation to 12 months post-operation: Scores were normalized with 50 equal to the national norm and 40 equal to one standard deviation below the norm, so a 12 month difference of 10 would equal a 1 standard deviation change; An increase is better.
Time Frame: 12 months
Population: Patients with 12 month completion of the SF12
Measure: Mean (Standard Deviation); unit: Normalized scores
Arm/Group | Flex HD | Strattice
Number analyzed (Participants) | 15 | 10
Normalized scores | 3 (8) | 2 (8)

10. Primary Outcome: Change in SF12 Mental Component Score Between Pre-operation and 12 Months Post-operation
Description: Change in SF12 Mental Component Score from pre-operation to 12 months post-operation: Scores were normalized with 50 equal to the national norm and 40 equal to one standard deviation below the norm; An increase is better.
Time Frame: 12 months
Population: Patients with 12 month completion of the SF12
Measure: Mean (Standard Deviation); unit: Normalized scores
Arm/Group | Flex HD | Strattice
Number analyzed (Participants) | 15 | 10
Normalized scores | 0 (12) | 6 (13)

ADVERSE EVENTS:
Time Frame: 24 Months
Groups:
- Strattice: Use of a second mesh type
  Strattice: Strattice mash for hernia repair
Arm/Group | Flex HD | Strattice
Serious Adverse Events (participants affected / at risk) | 0/18 | 2/17
Other Adverse Events (participants affected / at risk) | 14/18 | 14/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flex HD (N=18) | Strattice (N=17)
Abdominal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal Wound/Mesh Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flex HD (N=18) | Strattice (N=17)
Abdominal Abscess (Infections and infestations) | 2 (2) | 2 (2)
Abdominal Wound Infection (Infections and infestations) | 3 (3) | 2 (2)
Wound Infection (Infections and infestations) | 2 (2) | 3 (3)
Seroma (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) — Renal decompensation requiring dialysis
Abdominal Compartment Syndrome (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chronic Seroma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hernia Recurrence (Surgical and medical procedures) | 1 (1) | 2 (2)
Parastomal Hernia (Surgical and medical procedures) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This is a Prospective Quasi-experimental study. Patients were randomized in the traditional sense.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No